CLINICAL TRIAL: NCT03384134
Title: Mobile Technology to Improve Pain and Symptoms in Children With Cancer
Brief Title: Treating Pain in Children With Cancer: Pain Buddy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michelle Fortier, Study Principal Investigator, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20195027; 1R01CA222012-01 (NIH)
Record Dates: First submitted 2017-11-30; First posted 2017-12-27 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2024-09

CONDITIONS: Cancer
Keywords: cancer; cognitive and behavioral skills training intervention; pain; symptoms; quality of life
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: Following informed consent, participants will be randomized to the intervention or control group using a blocked randomization scheme with block size equal to 4 and stratified by age group, gender and diagnosis. An online program to will be used to derive an assignment. Patients will be randomized at a 1:1 ratio with equal numbers randomized to the intervention and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Buddy (Experimental): Children in this condition will continue with the care that has been prescribed for cancer- and chemotherapy-related pain and symptoms, which may include medications, medical visits, physical interventions, etc. Participants in this condition will complete daily diaries using Pain Buddy and will also be taught cognitive and behavioral coping skills, like deep breathing, imagery, and relaxation, to deal with pain and symptoms. The skills will be taught through the electronic tablet. Pain and symptom information, collected daily by Pain Buddy, will be sent to a health care provider on the oncology treatment team, who will contact patients when certain thresholds are reached and will instruct the patients on best ways to control pain and symptoms.
  Interventions: Other: Pain Buddy
- Control (No Intervention): Children in this condition will continue with the care that has been prescribed for cancer- and chemotherapy-related pain and symptoms, which may include medications, medical visits, physical interventions, etc. Participants in this condition will complete daily pain diaries using Pain Buddy, but will not receive skills training or remote monitoring of data.

INTERVENTIONS:
Other: Pain Buddy — Pain Buddy is a user interface (application) which contains a personalized avatar (Pain Buddy) to guide children and parents through daily diary entries using mobile devices. The Pain Buddy application has been designed to be used with children age 8-18, receiving outpatient chemotherapy, as well as their parents. Pain Buddy will capture real time pain data from patients and that will ultimately allow for remote monitoring of patient symptoms. Remote symptom monitoring in real time will provide an opportunity for implementation of appropriate interventions, thereby introducing the potential to decrease pain and symptoms and improve quality of life in children with cancer. The use of symptom monitoring and skills training will further increase patient engagement in healthcare.
  Arms: Pain Buddy

SUMMARY:
The purpose of this study is to examine the feasibility of the ambulatory monitoring protocol, called Pain Buddy, in documenting children's pain, symptoms and quality of life while receiving outpatient chemotherapy. The long term goal of Pain Buddy is to help doctors, nurses, and parents get the information they need to give children treatments for pain and symptom management that work. Using Pain Buddy, we aim to quantify the prevalence and intensity of daily pain and symptom episodes in children at home, data that will be used to develop a psychosocial intervention to be delivered electronically to children at home with a goal of improving quality of life. Secondary aims also include examining children's quality of life pre- and post- Pain Buddy and satisfaction with the use of Pain Buddy. This project has the potential to improve the quality of life of tens of thousands of children suffering from cancer each year using transformative mobile health information technology based approach to pain assessment and management.

DETAILED DESCRIPTION:
Approximately 12,000 children are diagnosed with cancer in the United States each year and the majority of these children will experience moderate to severe pain and disabling symptoms such as fatigue and nausea during the course of their illness. Survivors of childhood cancer are also at high-risk for long-term chronic pain. Unfortunately, the World Health Organization (WHO) indicates that current efforts to manage pain in pediatric oncology patients are seriously inadequate. Reasons for under treatment of pain and symptoms in children diagnosed with cancer are complex and are likely related to deficits in the process of assessment and management as well as lack of timely access to pharmacological and non-pharmacological interventions. Management of pain in this population is also compounded by the fact that increasing numbers of children currently receive chemotherapy on an outpatient basis due to advances in healthcare and changes in the medical-economical environment.

To date, interventions targeting pain and symptom management in the home setting of children suffering from cancer are seriously lacking. To address this significant gap, the candidate is proposing significant training in pediatric cancer pain and symptom management and an innovative two-phase research strategy. The first phase of research will focus on the development and formative evaluation of an innovative handheld electronic program (Pain Buddy) that provides remote monitoring of pain and symptoms and delivery of cognitive and behavioral skills training to children undergoing treatment for cancer. The second phase of this application involves evaluation of the efficacy of the program using a randomized controlled trial design. Pain Buddy will allow for collection of "real time" pain and symptom data that will be transmitted immediately and monitored remotely by the oncology treatment team. Remote symptom monitoring in real time will provide an opportunity for timely implementation of appropriate interventions, thereby introducing the potential to decrease pain and symptoms and improve quality of life. Pain Buddy will also deliver psychosocial skills training, teaching cognitive and behavioral strategies to manage pain and symptom-related distress. The skills training will target coping and self-efficacy in children without the need for face-to-face intervention which is not feasible in the majority of settings. Symptom monitoring and skills training will further increase patient engagement in their own health care, which is a main goal of the Institute of Medicine and many other organizations. The objectives outlined above will be accomplished by the following specific aims:

PHASE I: Development and Formative Evaluation Specific Aim 1: Through collaboration with the California Institute for Telecommunications and Information Technology (Calit2), develop and examine the usability of a cognitive and behavioral skills training intervention (Pain Buddy) delivered via electronic, handheld technology in conjunction with a validated pain and symptom assessment protocol (Jacob, E.) that will allow for monitoring of and response to pain and symptoms of pediatric oncology patients in real time.

Hypothesis 1. Children and their parents will demonstrate the ability to use Pain Buddy on the electronic device and will rate high levels of acceptability, usability and satisfaction on beta testing.

PHASE II: Randomized Controlled Trial of Pain Buddy Specific Aim 2: Using a randomized controlled trial design, we will examine the efficacy of Pain Buddy in managing pain and symptoms in children suffering from cancer.

Hypothesis 2. Children enrolled in the Pain Buddy group will report lower symptom-related distress as measured by the Memorial Symptom Assessment Scale (MSAS), compared to children in the monitoring group (primary outcome).

Hypothesis 3. Children in the Pain Buddy group will evidence lower pain severity and higher quality of life compared with children in the monitoring group (secondary outcomes).

Hypothesis 4. Children and nurses will demonstrate high rates of compliance (85% or greater) with Pain Buddy (secondary outcome).

The long-term goals of this research are to develop a usable, engaging electronic decision-support pain and symptom management intervention for children receiving outpatient chemotherapy using Smartphone technology and to examine the efficacy of the electronic decision-support intervention on children's pain and quality of life. These long-term goals will be accomplished through assessment of the data collected from patients, parents and physicians using the ambulatory monitoring protocol.

PHASE III: Multi-Site Randomized Controlled Trial of Pain Buddy

Primary Aim: Determine if Pain Buddy is more effective than attention control in reducing pain severity among children ages 8-18 years old undergoing outpatient cancer treatment.

Secondary Aims:

1. Examine the impact of Pain Buddy on symptom-related distress, health-related quality of life, functional status, and satisfaction with treatment experience.
2. Determine whether baseline characteristics of children (emotional functioning) and parents (stress, attitudes regarding analgesic use for children) moderate the effect of Pain Buddy on pain severity.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8-18 years
* Currently undergoing outpatient treatment for cancer
* Patients who are able to speak, read, and write in English. Parents who are able to speak, read, and write in English or Spanish
* Have home internet access to use Pain Buddy (the internet will be used to securely send the pain information to the research team).

Exclusion Criteria:

* Cognitive impairment, such as a developmental delay or mental retardation that would prevent children from being able to use the Pain Buddy program.
* Children diagnosed with acute myelogenous leukemia (AML) or acute promyelocytic leukemia (APL) as the treatment protocols for these children are largely inpatient, precluding use of the intervention.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 206 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in prevalence and intensity of pain episodes and other distressing physical and psychological symptoms. | Baseline and day 60
  As part of the daily electronic Pain Buddy diary, children are administered the Memorial Symptoms Assessment Scale. Children 8-9 receive an 8-item instrument and are asked to report frequency (i.e. a very short time, a medium amount, almost all the time) severity (i.e. a little, a medium amount, very), and how distressful (i.e. not at all, a little, a medium amount, very) each symptom was. Children 10-18 receive a 30-item instrument and are asked to report how often (i.e. almost never, sometimes, a lot, almost always), how severe (i.e. slight, moderate, severe, very severe), and how distressful (i.e. not at all, a little bit, somewhat, quite a bit, very much) each symptom was.
Changes in pain severity, location, and affective dimensions | Baseline and day 60
  Child's pain is assessed using the 3 components of the Adolescent Pediatric Pain Tool. 1. Children use a body outline/map to identify areas they are experiencing pain. 2. Children report pain intensity from "not in pain" (score of 0) and "worst pain" (score of 100) using the 100-mm Visual Analog Scale for Pain. 3. Children are presented with a pain quality word descriptor list within 4 categories (Sensory, affective, evaluative, and temporal).
Changes in children's quality of life since using Pain Buddy is assessed using the Pediatric Quality of Life Inventory (child self-report, ages 8-12, 13-18; parent report child ages 8-12, 13-18) | Baseline, day 60, and day 180
  Children and parents are asked to report on the child's health related quality of life. The measure incorporates a generic, cancer, and fatigue module and asks question on a 5-point likert scale from 0 ("Never") to 4 ("Almost Always") For questions like "I have trouble sleeping." Higher scores on the scale suggest a better health related quality of life. These responses are useful in understanding pain information collected in Pain Buddy.
Changes in Children's Anxiety and Depression assessed using the Revised Child Anxiety and Depression Scale (RCADS) | Baseline, day 60, and day 180
  Parent and Child's self report on 47-item scale with subscales including separation anxiety, social phobia, generalized anxiety, panic disorder, obsessive compulsive disorder, and major depression. Items are rated on a 4-point Likert scale from 0 ("never") to 3 ("always"). Higher scores suggest higher levels of anxiety and depression.
State-Trait Anxiety Inventory (STAI) (parent self-report) | Baseline
  Only the Trait section of the questionnaire is administered to parents to assess their self reported anxiety. Items rated on a 4-point Likert Scale from 1 ("Almost Never") to 4 ("Almost Always"). Higher scores suggest higher levels of anxiety.
Changes in Perceived Stress (parent self-report) | Baseline, day 60, and day 180
  Parents are administered the 14-item Perceived Stress Scale and asked to rate statements such as "In the past month, how often have you been upset because of something that happened unexpectedly?" and "In the past month how often have you felt that things were going your way?" Subjects rate the items on a 5-point Likert-type scale with higher scores reflecting greater perceived stress.
Medication Attitude Questionnaire (MAQ) (parent self-report) | Baseline
  Parents were asked to report their attitudes regarding use of pain medication for treating children's pain. The factors assessed were Appropriate-Use (e.g., "Giving children pain medication for pain teaches proper use of drugs"), Side-Effects (e.g., "Side effects are something to worry about when giving children pain medication"), and Avoidance (e.g., "Pain medication works best if saved for when the pain is quite bad").

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Fortier, Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No